CLINICAL TRIAL: NCT05226923
Title: A Phase 1 Randomized, Double-Blind, Placebo-Controlled, Dose-Escalation Study to Assess the Safety, Tolerability, and Pharmacokinetics of Single and Repeat Doses of KSP-1007 Alone and Coadministered With Meropenem in Healthy Subjects
Brief Title: Study of the Safety and Pharmacokinetics of KSP-1007 Alone and Coadministered With Meropenem in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sumitovant Biopharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: KSP-1007-101
Record Dates: First submitted 2022-01-07; First posted 2022-02-07 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Bacterial Infections
Keywords: Bacterial Disease; Bacterial Infection; Bacterial Infections; Bacterial; Healthy Volunteers
MeSH Terms: conditions — Bacterial Infections | interventions — Meropenem

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- KSP-1007 single ascending dose (Experimental): Single, ascending intravenous dose of KSP-1007
  Interventions: Drug: KSP-1007
- Placebo single dose (Placebo Comparator): Single dose of placebo (0.9% normal saline)
  Interventions: Other: Placebo:0.9% sodium chloride
- KSP-1007 multiple ascending dose (Experimental): Multiple, ascending, intravenous doses of KSP-1007
  Interventions: Drug: KSP-1007
- Placebo multiple dose (Placebo Comparator): Multiple doses of placebo (0.9% saline)
  Interventions: Other: Placebo:0.9% sodium chloride
- KSP-1007 multiple ascending dose + Meropenem multiple dose (Experimental): Multiple, ascending intravenous doses of KSP-1007 and multiple doses of meropenem (fixed dose)
  Interventions: Drug: KSP-1007; Drug: Meropenem
- Placebo + Meropenem multiple dose (Placebo Comparator): Multiple doses of placebo (0.9% normal saline) plus multiple doses of meropenem (fixed dose)
  Interventions: Other: Placebo:0.9% sodium chloride; Drug: Meropenem

INTERVENTIONS:
Drug: KSP-1007 — Single and multiple doses, intravenous administration
  Arms: KSP-1007 multiple ascending dose; KSP-1007 multiple ascending dose + Meropenem multiple dose; KSP-1007 single ascending dose
Other: Placebo:0.9% sodium chloride — Single and multiple doses, intravenous administration
  Arms: Placebo + Meropenem multiple dose; Placebo multiple dose; Placebo single dose
Drug: Meropenem — Multiple doses, intravenous administration
  Arms: KSP-1007 multiple ascending dose + Meropenem multiple dose; Placebo + Meropenem multiple dose

SUMMARY:
This study is a first-in-human, Phase 1, randomized, double- blind, four-part, dose-escalation study to assess the safety, tolerability, and pharmacokinetics of single (Part 1) and repeat (Part 2) escalating intravenous doses of KSP-1007. Repeated escalating doses of KSP-1007 will be co-administered with meropenem (Part 3) and single, ascending doses of KSP-1007 will be administered alone in healthy Japanese subjects (Part 4)

DETAILED DESCRIPTION:
Carbapenem-resistant Gram-negative bacteria are responsible for serious, life-threatening infections and are regarded as an urgent threat by the Centers for Disease Control and Prevention and the World Health Organizations. One principal mechanism of carbapenem resistance is bacterial production of carbapenemases, which reduce the effectiveness of meropenem and other carbapenem class antibiotics. Sumitovant Biopharma is developing a fixed combination of meropenem and KSP-1007 for the treatment of serious bacterial infections.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects 18 to 55 years of age, inclusive
* Females that engage in heterosexual activity must agree to use a highly selective birth control (BC) method (< 1% failure rate per year) throughout the study, or have a documented reproductive status of non-childbearing based on medical history, or is postmenopausal
* Males that engage in heterosexual activity that has the risk of pregnancy must agree to use effective BC and agree to not donate sperm during the study and for at least 90 days after the last dose of the study medication
* Body mass index (BMI) 2: 18 kg/m2 and :s 32 kg/m2

Exclusion Criteria:

* History of Gilbert's Syndrome
* History of severe allergic reactions to β-lactams or β-lactamase inhibitors or a history allergic reactions to multiple medications.
* Pregnant female, determined by positive serum or urine human chorionic gonadotropin pregnancy test at Screening, or prior to dosing
* Lactating female
* Donation of plasma within 7 days prior to dosing. Donation or loss of blood (excluding volume drawn at Screening) of > 499 mL within 56 days prior to Day 1
* Participation in a study with an investigational drug or device study with last dose of investigational drug within 30 days (90 days if the study involved a biologic, cellular, or vaccine product) or 5 half-lives, whichever is longer, before study treatment administration
* Subjects with abnormal hepatic and/or renal function, that could interfere with the metabolism, and/or excretion of the study treatments
* Abnormal blood pressure, either low (defined as < 90 mmHg systolic and/ or < 45 mmHg diastolic) or high (defined as > 140 mmHg systolic and/ or > 90 mmHg diastolic) at Screening
* Positive serology for hepatitis B virus (HBV), hepatitis C virus (HCV), or HIV at Screening. Subjects who test positive for hepatitis B core antibody (HBcAb) or hepatitis B surface antigen (HBsAg) also will be ineligible. Evidence of prior HBV vaccination (positive hepatitis B surface antibody [HBsAb)) is not exclusionary.
* Subjects unable to abstain from alcohol for 48 hours prior to admission through to completion of the Follow-up visit

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 123 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events assessed by subject . | up to Day 14
  Incidence of adverse events

SECONDARY OUTCOMES:
Peak plasma concentration of KSP-1007 | Up to 5 days after dosing
  The plasma concentration of KSP-1007 will be measured over time, and the peak plasma concentration, or Cmax, of KSP-1007 will be determined
Plasma concentration of KSP-1007 versus time curve | Up to 5 days after dosing
  The plasma concentration of KSP-1007 will be measured over time and the area under the curve, or AUC, of KSP-1007 will be determined
Cumulative amount of KSP-1007 excreted in urine over time | Up to 5 days after start of dosing
  Total amount of unchanged drug excreted in urine over a dosing interval
Renal clearance of KSP-1007 in urine over time | Up to 5 days after start of dosing
  Renal clearance in urine. Urine was collected up to 5 days after dosing.
Peak plasma concentration of meropenem | Up to 5 days after start of dosing
  The plasma concentration of meropenem will be measured over time, and the peak plasma concentration, or Cmax, of meropenem will be determined
Plasma concentration versus time curve of meropenem | Up to 5 days after start of dosing
  The plasma concentration of meropenem will be measured over time and the area under the curve, or AUC, of meropenem will be determined
Cumulative amount of meropenem excreted in urine over time | Up to 5 days after start of dosing
  Total amount of unchanged drug excreted in urine over a dosing interval.
Renal clearance of meropenem in urine over time | Up to 5 days after start of dosing
  Renal clearance in urine. Urine was collected up to 5 days after dosing.
ECG QTcF interval | 24 hours after start of dosing
  Change from baseline QTcF interval

CONTACTS AND LOCATIONS:
Overall Officials: Hayes Dansky, M.D., Study Director — Sumitovant Biopharma, Inc.
Locations (1):
- PRA Health Sciences, Lenexa, Kansas, United States

IPD SHARING:
Plan to Share IPD: No